CLINICAL TRIAL: NCT06430983
Title: Recurrent Liver Cancer: Reconceptualization and Reevaluation
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yewei Zhang, Chief Physician, Nanjing Medical University
Other Study IDs: 2024KY16401
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Liver Cancer; Primary Liver Cancer
Keywords: Recurrent Liver Cancer; Primary Liver Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Training Set for Recurrent Liver Cancer Patient: The training set for recurrent liver cancer patients is a subset of data collected from individuals who have been diagnosed with liver cancer that has returned after a period of remission or initial treatment. This data set is used to train machine learning models or other statistical methods to identify patterns or biomarkers that are indicative of cancer recurrence. The training set typically includes information such as patient demographics, medical history, previous treatments, and biological data, such as genetic mutations, protein levels, or imaging results. The goal is to use this data to develop a model that can accurately predict the recurrence of liver cancer in other patients, which can then be validated and tested using a separate data set, known as the validation set.
- Validation Set for Recurrent Liver Cancer Patient: The validation set for recurrent liver cancer patients is a distinct subset of data that is used to assess the performance and generalizability of a model or hypothesis developed from a training set. This set includes data from patients with recurrent liver cancer who were not part of the original training set. The purpose of the validation set is to test the model's ability to accurately predict or classify cases of recurrent liver cancer in a population that it has not been exposed to during its training phase.

SUMMARY:
The goal of this observational study is to determine if a specific protein can serve as a novel indicator for the recurrence of liver cancer. The study will focus on recurrent liver cancer patients and compare participants to primary liver cancer patients as controls. The primary purpose is to assess whether the elevated levels of this protein can be used to monitor the recurrence of liver cancer.

The main questions it aims to answer are:

Is the levels of the protein significantly elevated in recurrent liver cancer patients compared to primary liver cancer patients? Can the protein be used as a reliable biomarker for the early detection of liver cancer recurrence?

Researchers will compare the protein levels in the following groups:

50 recurrent liver cancer patients (training set) with abnormally high levels of the protein.

250 recurrent liver cancer patients (validation set) to confirm the protein's elevation in a separate cohort.

Participants will be required to:

* Provide blood samples for protein analysis.
* Undergo regular follow-up visits for monitoring and data collection.
* Allow access to their medical records for relevant clinical information.

DETAILED DESCRIPTION:
As part of the patient registry, investigators will implement the following registration procedures and other quality factors:

Screening and Recruitment: Eligible patients will be screened and recruited through hospital liver cancer outpatient clinics and wards. Patients must meet the diagnostic criteria for recurrent or primary liver cancer and be willing to participate in the study.

Data Collection: Clinical information of participants will be collected, including demographic characteristics, medical history, treatment regimens, and follow-up outcomes. Data will be entered and verified by professionals to ensure accuracy and completeness.

Quality Control: Strict quality control measures will be implemented, including data audits, sample management, and laboratory testing. Regular reviews and validations of the data will be conducted to ensure the reliability and replicability of the study results.

Data Security: The privacy and personal information of participants will be protected. All data will be stored in a secure environment and comply with relevant laws, regulations, and ethical guidelines.

Ethical Review: The research protocol has been approved by the ethics committee, ensuring that the conduct of the study meets ethical standards and the protection of patient rights.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary hepatocellular carcinoma or diagnosed with non-HCC
* The patient or the patient's legal representative must be able to read, understand, and sign the informed consent form
* Agree to provide blood samples and have good clinical compliance
* Complete clinical basic information, including: the patient's unique traceability number (ID card number/outpatient number/health insurance card number), age, gender, imaging and/or pathological diagnosis results (for patients with primary liver disease), imaging examination confirmed heteromorphic liver cancer (for non-HCC patients)

Exclusion Criteria:

* Pregnant women
* Those who have received organ transplantation
* Non-HCC patients diagnosed with other tumors
* Patients with primary hepatocellular carcinoma complicated by other tumors
* Those judged by the researcher as not meeting the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with primary hepatocellular carcinoma (HCC) and non-HCC liver cancers. Inclusion criteria are: diagnosis of primary HCC or non-HCC, ability to provide informed consent, agreement to supply blood samples, and clinical data completeness. Exclusion criteria include pregnancy, organ transplantation, other tumor diagnoses in non-HCC patients, HCC with other tumors, and researcher-determined ineligibility. The sample size is limited to ensure data precision and study validity.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Novel Protein Indicator | Assessed at the end of the study (up to 3 years), once all patient data has been collected and analyzed.
  The primary outcome is to determine the sensitivity and specificity of the novel protein indicator in predicting the recurrence of liver cancer. This will be assessed by constructing a Receiver Operating Characteristic (ROC) curve and establishing a threshold value that maximizes the true positive rate (sensitivity) and minimizes the false positive rate (1-specificity). The ROC curve will visually represent the trade-off between sensitivity and specificity for different threshold values.
Positive and Negative Predictive Values | Calculated after the threshold value has been determined and applied to the patient data (up to 3 years).
  The secondary outcome is to calculate the positive predictive value (PPV) and negative predictive value (NPV) of the novel protein indicator. The PPV represents the probability that patients with an elevated indicator level will experience cancer recurrence, while the NPV represents the probability that patients with a non-elevated indicator level will remain free of recurrence. These values will provide insight into the clinical utility of the indicator.

SECONDARY OUTCOMES:
Overall Survival (OS) | Monitored throughout the study and reported at 1 year, 2 years, and study completion (up to 5 years).
  Overall survival (OS) is a critical endpoint that measures the length of time from the start of the study until the death of a patient. It provides an assessment of the long-term outcome for patients with liver cancer and will be used to evaluate the prognostic value of the novel protein indicator.
Progression-Free Survival (PFS) | Assessed at each follow-up visit, every 3 months for the first 2 years, then every 6 months until study completion (up to 5 years).
  Progression-free survival (PFS) is the length of time during and after the treatment of a disease that a patient lives without the disease getting worse. In the context of this study, PFS will be used to measure the time from study entry until the cancer progresses or the patient dies from any cause, providing an intermediate endpoint that reflects the control of disease progression.
Disease-Free Survival (DFS) | Monitored and reported at 6 months, 1 year, 2 years, and study completion (up to 5 years).
  Disease-free survival (DFS) is the period after treatment during which there is no evidence of active cancer. It is a measure of the effectiveness of treatment in eliminating cancer cells. DFS will be calculated from the time of treatment initiation until the first sign of cancer recurrence or the end of the study.
Time to Progression (TTP) | Measured from the initiation of the study intervention until progression or defined worsening, assessed at each follow-up visit (every 3 months for the first 2 years, then every 6 months until study completion, up to 5 years).
  Time to progression (TTP) is the interval from the start of treatment until the tumor progresses or the patient's condition worsens to a defined level. This endpoint is particularly relevant for evaluating the effectiveness of the novel protein indicator in predicting and monitoring disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: zhang yewei, doctor, Study Chair — Nanjing Medical University
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China